CLINICAL TRIAL: NCT04323280
Title: Dexamethasone Compared to Non-steroidal Anti-inflammatory Drugs in the Treatment of Acute Pericarditis: a Non-inferiority Randomized Controlled Trial (Dexa-P)
Brief Title: Dexamethasone Compared to Non-steroidal Anti-inflammatory Drugs in the Treatment of Acute Pericarditis
Acronym: Dexa-P
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in enrollment of patients
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-0543-19
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Pericarditis Acute
Keywords: Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomised, non-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Active Comparator): Ibuprofen 600mg every 8 hours for one week followed by tapering of dose by 200mg every week (3 weeks of therapy), in addition to Colchicine 0.5mg daily (<70kg) or 0.5mg twice daily (>70kg) for 3 months
  Interventions: Drug: NSAID therapy
- Dexamethasone therapy (Experimental): Dexamethasone therapy 20 mg once daily per os for 4 day in addition to colchicine therapy for 3 months 0.5mg daily (<70kg) or 0.5mg twice daily (>70kg)
  Interventions: Drug: Dexamethasone therapy

INTERVENTIONS:
Drug: Dexamethasone therapy — Dexamethasone 20MG once daily for 4 days with additional colchicine therapy for 3 months
  Arms: Dexamethasone therapy
Drug: NSAID therapy — NSAIDS (Ibuprofen or Aspirin) or Glucocorticoid (Prednisone) therapy for 3 weeks with addional colchicine therapy for 3 months
  Arms: Conventional Therapy

SUMMARY:
The treatment of acute pericarditis is empiric and is based on treatment with medications with anti-inflammatory properties such as non-steroidal anti-inflammatory drugs (NSAID) and corticosteroids. However, this therapy is given as a relatively long course of therapy (≥ 3 weeks) and can be associated with substantial side effects.

Dexamethasone is a potent corticosteroid that has not been investigated an alternative to conventional therapy in patients with acute pericarditis.

Dexamethasone is an inexpensive drug and can be given in an oral tablet form. It has a quick onset of action, relatively long duration of action and is therefore often given in high doses for short periods.

Dexamethasone has been shown to be a safe therapeutic option in ITP (Immune Thrombocytopenia), another disease in which steroids are an accepted treatment option. The abundant data on using dexamethasone in comparison to longer prednisone-based regimens has been evaluated in this disease and has shown to be effective and without the longer exposure time to steroids and potential side effects. This data shows that dexamethasone can be a safe therapeutic option.

The investigators hypothesize that therapy with short term, high dose dexamethasone will offer better clinical responses to NSAID therapy in the treatment of acute pericarditis with less potential side effects compared to NSAID therapy.

The Investigators aim to conduct a randomised, non-blinded trial assessing the use of dexamethasone as an alternative to NSAID for use in patients with acute pericarditis.

DETAILED DESCRIPTION:
Dexamethasone compared to Non-steroidal anti-inflammatory drugs in the treatment of acute pericarditis: a non-inferiority randomized controlled trial (Dexa-P)

Objectives:

The investigators hypothesize that therapy with short term, high dose dexamethasone will offer better clinical responses to NSAID therapy with less potential side effects compared to conventional therapy

Trial design:

A randomised, non-blinded trial assessing the use of dexamethasone as an alternative to NSAID therapy for use in patients with acute pericarditis.

Quality Assurance:

After the first 3 participants have been enrolled and completed a month of follow up, the preliminary findings will be forwarded to the quality control committee of the Helsinki Ethics Committee of Rabin Medical Center

Withdrawal of participants:

Participants are free to discontinue their participation in the study at any time and without prejudice to further treatment.

A participant may withdraw or be withdrawn from the study for the following reasons:

* Subject withdrew consent.
* Severe Adverse Event (As described below) Reasons for withdrawal will be documented. In cases of more than one reason for early withdrawal from the study, the most significant reason will be stated.

Replacement of withdrawn participants:

Withdrawn randomized participants will not be replaced.

Discontinuing or modifying allocated interventions:

If a participant has incessant pericarditis within one month of therapy:

* Participants in the dexamethasone arm will be given another cycle of dexamethasone therapy of 20mg for 4 days can be given. If there is a further persistence, prednisone therapy will then be initiated.
* Participants in the NSAID therapy arm will be changes to prednisone therapy

Definition of incessant pericarditis:

Recurrence of pleuritic chest pain and one or more of the following signs:

1. Pericardial friction rub
2. Electrocardiographic changes specific to pericarditis (concave ST elevation, PR depression)
3. Echocardiographic evidence of pericardial effusion

3) An elevation in inflammatory markers (white-cell count, or C-reactive protein level) without a symptom-free interval of 6 weeks or longer after the first acute event.

If participant is hospitalized with a possible side effect, the treating physician will be notified to assess for modifying the participant allocation.

Concomitant care:

There are no prohibited concomitant medications. Participants should continue to take drugs for other co-morbidities as usual.

Participant Timeline:

The enrollment will be done within 72 hours of initial assessment. Each participant will undergo eligibility screen and suitable participants will receive informed consent. The allocation will be determined immediately after the participant will be found to be eligible and will be made randomly.

Once participants are identified with an initial episode of acute pericarditis and informed consent is given, an initial assessment will be done.

This will include baseline blood tests - including baseline liver and renal function tests, full blood count and C-reactive protein.

All participants will undergo echocardiographic imaging at baseline. There are two possible interventions: dexamethasone therapy or NSAID therapy. Participants will be followed up at 1 weeks, 1 month, 6 months and 12 months after treatment initiation.

The follow up will be telephonically at 1 week, 6 months and 12 months. At the 1 month follow up, clinical assessment, inflammatory marker and a repeat echocardiogram will be performed. A repeat echocardiogram will be performed at 12 months. This follow up will be at the pericardial disease clinic at Rabin Medical Center

Sample size:

Assuming a success rate 85% in the NSAIDS group and 87% in the Dexamethasone intervention group, with a margin of non-inferiority of 10%, the sample size calculated was 208. (Alpha = 0.05, beta=0.2). Noninferiority would be shown if the upper boundary of the 95% confidence interval was 10 percentage points or less. A 10 percentage-point noninferiority margin was considered to be an acceptable difference in recurrence rate.

Recruitment:

Investigators will include physicians in the emergency room and admission setting to help identify and recruit participants.

Methods: Data Collection, management and analysis

Enrollment:

First assessment including baseline variables and suitability of the participant to the study will be made during the enrollment, by the study coordinators.

In addition demographic and clinical characteristics will be recorded. The data will be collected during an interview of the participant or with assistance of the computerized medical records.

Furthermore, laboratory tests such as blood count, liver and kidneys functions and C reactive protein will be made and be recorded for each participant.

Interventions:

The type of intervention will be recorded by the study coordinators for each participant according to the allocation group.

Assessments of outcomes:

The primary outcome at each follow up, both telephonically and on clinical follow up The secondary outcomes will be assessed telephonically and using the medical computerized systems.

Data management:

All data regarding the participant's hospitalization: Baselines variables, interventions and glucose levels will be stored in secured excel documents for each study group.

Data regarding the participant's outcomes will be stored in a different secured excel documents for each study group.

The coding of the documents and the separation between the hospitalization and follow up period data is designated to ensure the investigator blinding.

Statistical analysis:

The primary outcome is the occurrence of Recurrent Pericarditis within 12 months. This will be calculated by bivariate analysis as relative risk. The secondary outcome of time to recurrence will be plotted using Kaplan-Meier curves and compared using the Log-rank test (unadjusted analysis), Hazard ratio for the risk of the primary analysis between the control and Dexamethasone arm will be calculated using a univariate cox proportional hazards ratio model (unadjusted analysis). Further secondary outcomes will be analysed by bivariate analysis.

Methods: monitoring Harms: Side effects will be monitoring during therapy as defined

ELIGIBILITY:
Inclusion Criteria:

* Patient with first presentation of acute pericarditis (both idiopathic and post pericardiectomy)
* Patients diagnosed according to accepted clinical findings: 2 of the 4 following criteria: chest pain, pericardial friction rub, ECG changes typical for pericarditis and/or pericardial effusion.
* Patients over the age of 18 years

Exclusion Criteria:

* Patient with Uncontrolled Diabetes (as defined as hyperglycaemia >300mg/dl at presentation or HBA1C>9% (if known))
* Patients with a known allergy to steroid therapy
* Patient with a known allergy to NSAID therapy
* Patients with a known contraindication to colchicine therapy
* Pregnancy or lactating women
* Patients with systemic fungal infection
* Patients with a known pericardial effusion of tuberculous, purulent, or neoplastic causes
* Patients with chronic steroid use
* Patients with a known rheumatological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Occurrence of Recurrent Pericarditis within 12 months | 12 months
  Definition of Recurrent Pericarditis:
  Recurrence of pleuritic chest pain and one or more of the following signs:
  1. Pericardial friction rub
  2. Electrocardiographic changes specific to pericarditis (concave ST elevation, PR depression)
  3. Echocardiographic evidence of pericardial effusion
  4. An elevation in inflammatory markers (white-cell count,or C-reactive protein level) with a symptom-free interval of 6 weeks or longer after the first acute event.

SECONDARY OUTCOMES:
The time to first recurrence | 12 months
  Average number of days to first recurrence of pericarditis (as per definition above) in each arm
Disease-related re-hospitalization | 12 months
  Number of participants in each arm that are hospitalization due to recurrent pericarditis
Occurrence of new onset Atrial Fibrillation | 12 months
  Incidence of new onset atrial fibrillation in each arm
Cardiac Tamponade | 1 month
  Number of participants that develop cardiac tamponade in each arm
Constrictive Pericarditis | 12 months
  Number of participants that develop constrictive pericarditis in each arm
Side effects during therapy | During therapy (4 days or 3 weeks depending on arm of therapy)
  Number of Participants in each arm that experience:
  * Gastrointestinal Disorder during therapy : diarrhoea (>3 times in 24 hours), vomiting (>3 times in 24 hours) due to therapy
  * Renal dysfunction (An increase in serum creatine >1.5 times baseline which has occurred within 1 week of therapy)
  * Hyperkalaemia during therapy (> 6 mEq/l)
  * Development of Severe Hypertension during therapy - Diastolic Blood Pressure >110mmHg
  * Hyperglycaemia during therapy >200mg/dl
  * Bleeding Event during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nili Schamroth Pravda, MbbCH, Study Chair — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No